CLINICAL TRIAL: NCT06842251
Title: A COMPARISON of EFFECT of TWO INSTRUMENTATION TECHNIQUES on the INCIDENCE of POST-ENDODONTIC PAIN in PATIENTS UNDERGOING ROOT CANAL TREATMENT
Brief Title: To COMPARE the EFFECT of TWO INSTRUMENTATION TECHNIQUES on the INCIDENCE of POST-ENDODONTIC PAIN in PATIENTS UNDERGOING ROOT CANAL TREATMENT in TEETH with IRREVERSIBLE PULPITIS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Urooj Fatima (Other)
Responsible Party: Sponsor-Investigator, Urooj Fatima, Post Graduate Trainee, Margalla Institute of Health Sciences
Organization: Margalla Institute of Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DU/249/24
Record Dates: First submitted 2025-02-07; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-09

CONDITIONS: Irreversible Pulpitis; Symptomatic Irreversible Pulpitis; Asymptomatic Irreversible Pulpitis
Keywords: Symptomatic Irreversible Pulpitis; Asymptomatic Irreversible Pulpitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A : Rotary Crown Down Technique (Active Comparator): patients undergoing root canal treatment with rotary crown down technique
  Interventions: Other: Rotary Crown Down Technique
- Group B : Manual Step Back Technique (Active Comparator): Patients undergoing root canal treatment with manual step back technique
  Interventions: Other: Manual Step Back Technique

INTERVENTIONS:
Other: Rotary Crown Down Technique — Root canal treatment with rotary instrument is done using crown down approach and post endodontic pain measured after 4,12,24,48 hours.
  Arms: Group A : Rotary Crown Down Technique
Other: Manual Step Back Technique — Root canal treatment with manual instruments using step back technique and post endodontic pain measured at 4,12,24,48 hours .
  Arms: Group B : Manual Step Back Technique

SUMMARY:
The aim of this study is to compare the post endodontic pain in patients presenting with irreversible pulpitis and undergoing root canal treatment with two techniques. One is rotary crown down technique and other is manual step back technique. Patients visiting OPD will be selected after fulfilment of inclusion criteria and randomly divided into two groups. In Group A rotary instrument with Crown Down approach is used and in Group B manual instrumentation with Step Back technique is used. Post endodontic pain will be graded using VAS scale at 4,12,24 and 48 hours.

DETAILED DESCRIPTION:
The main objective of this study was to compare the effect of step back manual and crown down rotary techniques on post endodontic pain in teeth with irreversible pulpitis after root canal treatment .Crown Down technique involves the preparation of the coronal portion of the root canal, followed by the middle and apical third of the root canal .Step Back technique involves initial apical preparation followed by step-wise coronal preparation to create tapers .By using WHO sample size calculator, sample size is 70 having 35 in each group.

Inclusion criteria include patients of both genders having age 18-70 years, no history of analgesics within the past 1 week, subjects with no periapical radiolucency, teeth having completely formed tooth apex, permanent posterior teeth with symptomatic/asymptomatic irreversible pulpitis, subjects who provided the consent for study participation. Exclusion criteria include subjects with a history of trauma, previous root canal treatment, associated systemic diseases, pregnant females ,subjects on analgesics or antibiotics ,complaints of tenderness and pain within the past 5 days, extreme root curvature, calcified canals, external or internal resorption. The study will be conducted after permission from institutional ethics review committee. Patients presenting in Operative outpatient department at Margalla Dental Hospital, Rawalpindi, and fulfilling inclusion criteria will be included in this study.

After ensuring the general health of patients by taking a medical history, the pulp and periapical status of the teeth will be assessed by thermal and electric tests, percussion, palpation, and radiography. The patients will then be briefed about the study, and written informed consent will be obtained from them. Local anesthesia will be administered by an inferior alveolar nerve block with the injection of 1.8 mL lidocaine plus 1:80,000 epinephrine. Optimal depth of anesthesia will be ensured by electric and thermal tests. After ensuring optimal depth of anesthesia, the access cavity will be prepared, and the orifices will be negotiated and canals will be instrumented by the crown down rotary or step down manual technique based on the group allocation of the teeth. The patients will not be aware of the technique used for their endodontic treatment. VAS scale will be used to grade the post endodontic pain at different time intervals after procedure at 4,12,24 and 48 hours. All data will be recorded in a specially designed Performa. Data will be entered in SPSS version 24. The data will be expressed in the means and standard deviations. Chi square will be applied and Independent sample t test will be used to evaluate difference in the mean age of the two groups. P < 0.05 will be considered statistically significant.

Local anesthesia will be administered by an inferior alveolar nerve block with the injection of 1.8 mL lidocaine plus 1:80,000 epinephrine. Optimal depth of anesthesia will be ensured by electric and thermal tests. After ensuring optimal depth of anesthesia, the access cavity will be prepared, and the orifices will be negotiated and canals will be instrumented by the crown down rotary or step down manual technique based on the group allocation of the teeth. The patients will not be aware of the technique used for their endodontic treatment. VAS scale will be used to grade the post endodontic pain at different time intervals after procedure at 4,12,24 and 48+ hours. All data will be recorded in a specially designed performa.Data will be entered in SPSS version 24. The data will be expressed in the means and standard deviations.Independent sample t test will be used to evaluate difference in the mean age of the two groups. P < 0.05 will be considered statistically significant.

Exclusion criteria include subjects with a history of trauma, previous root canal treatment ,associated systemic diseases ,pregnant females ,subjects on analgesics or antibiotics ,complaints of tenderness and pain within the past 5 days ,extreme root curvature, calcified canals ,external or internal resorption.

ELIGIBILITY:
Inclusion Criteria:1.Patients of both genders having age 18-70 years, no history of analgesics within the past 1 week ,subjects with no periapical radiolucency, teeth having completely formed tooth apex ,permanent posterior teeth with symptomatic/asymptomatic irreversible pulpitis, subjects who provided the consent for study participation

-

Exclusion Criteria: Subjects with a history of trauma, previous root canal treatment, associated systemic diseases ,pregnant females, subjects on analgesics or antibiotics, complaints of tenderness and pain within the past 5 days, extreme root curvature, calcified canals ,external or internal resorption.

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Post endodontic pain | 6 months
  post operative pain measured through visual analogue scale(VAS) from readings no pain 0, mid pain taken as 0-2, moderate as 2-5, severe taken as 5-10

CONTACTS AND LOCATIONS:
Overall Officials: Urooj Fatima, Post Graduate Trainee, Principal Investigator — Margalla Institute of Health Sciences
Locations (1):
- Margalla Institute of Health Sciences, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No